CLINICAL TRIAL: NCT03723837
Title: Cross-sectional Study to Assess Persistence of Immunity Conferred by a Single IPV Dose Administered in the Expanded Program on Immunization(EPI) Routine Immunization Schedule
Brief Title: Persistence of IPV Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Collaborators: World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Kumar Sharma, Co PI, Associate Professor, Department of Pediatrics, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69/2018
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Poliomyelitis
Keywords: IPV; Routine immunization; Single dose; Persistence of immunity
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm A (Active Comparator): Children {Age > 24 months and who received a single dose Inactivated Polio Vaccine (IPV) at the time of routine immunization} in this arm will receive an IPV (0.5ml) intramuscularly at the time of enrolment in the trial
  Interventions: Biological: Inactivated Polio Vaccine (IPV)
- Study arm B (Active Comparator): Children {Age 7-12 months and have not received any IPV till date of enrolment} in this arm will receive an Inactivated Polio Vaccine, IPV (0.5 ml) intramuscularly at the time of enrolment in the trial and a repeat dose of IPV (0.5 ml) after 1 month
  Interventions: Biological: Inactivated Polio Vaccine (IPV)

INTERVENTIONS:
Biological: Inactivated Polio Vaccine (IPV) — Children receive one or two doses of IPV based on study arm they fall in

SUMMARY:
In 2015, Strategic Advisory Group of Experts in Immunization (SAGE) recommended the global switch from trivalent to bivalent oral poliovirus vaccine (OPV) that does not contain type 2 poliovirus and introduction of a single dose of inactivated poliovirus vaccine (IPV) to maintain population immunity to type 2 polio to reduce the risk of vaccine derived polio. Following SAGE recommendations, Nepal introduced one dose of IPV in routine immunization in 2015 followed by withdrawal trivalent OPV in April 2016. However, Nepal, like many other countries had to stop vaccination by the end of 2016 because of a global shortage of IPV.

Single dose of IPV induces detectable antibodies in 34% to 80% of infants, compared to >90% after three doses and most of seronegative children (84-98%) are "immunologically primed" by the first dose. Primed individuals produce protective antibody levels in serum within one week of exposure to a new dose of IPV or OPV. However, it is unknown whether seroconversion or priming responses persist, and for how long they persist after the single dose of IPV. IPV immunogenicity for vaccine delivered low-resource countries may also be inferior to that observed in clinical trials because of program factors that decrease vaccine efficacy.

This cross sectional study aims to determine whether the immune response provided by a single dose of IPV delivered through routine immunization services persists for more than a year.

The study will be implemented in three study sites in Kathmandu, Nepal during November 2018- July 2019.

Information generated from this study is expected to allow better estimation of children partially protected (primed) or fully protected against type 2 poliovirus depending on coverage and time since last IPV vaccination. These estimates will help inform the Global Polio Eradication Initiative (GPEI) on vaccine choices for responding to type 2 vaccine derived poliovirus (VDPV) outbreaks and will help guide decisions on polio immunization schedules for Nepal and for other countries in future.

DETAILED DESCRIPTION:
Background and Rationale

Importance of Poliomyelitis and Polioviruses and vaccine

There are three polioviruses types, 1, 2 and 3, with minimal cross-immunity. About 1/200 infections (depending on the type of poliovirus) produce paralytic poliomyelitis. An estimated 5-10% of individuals with paralytic poliomyelitis die and the remaining suffer from lifelong paralysis of one or more limbs without a cure. The presence of detectable antibodies in blood against each type protects against paralytic poliomyelitis, but intestinal immunity develops only after exposure to live poliovirus (vaccine or wild). Oral poliovirus vaccines that contain attenuated poliovirus strains and inactivated poliovirus vaccine both induce humoral immunity and protect against paralysis. OPV can also immunize or boost immunity of close contacts through secondary spread and trivalent OPV (tOPV) with poliovirus types 1, 2 and 3, was the vaccine of choice for polio eradication.

The immunological response to poliovirus vaccines is evaluated by measuring type-specific poliovirus antibodies using neutralization assays and can be detected as early as 1 to 3 days after infection with WPV or receipt of OPV or IPV. Antibody titers usually decline in the first two years (10- to 100-fold reduction) and then plateau, persisting for many years. However, administration of additional doses of vaccine or new exposures to wild poliovirus, induces a quick rise in antibody titers, with a peak reached within one week after the dose due to induction of "priming" or immunological memory.

Changes in polio vaccine use with progress in global polio eradication

Global Polio Eradication Initiative (GPEI) reduced polio cases enormously with the use of the tOPV in routine immunization and campaigns and WPV circulation is now limited to a few areas of the world. However, problems related to vaccines emerged. OPV strains may occasionally cause paralysis in vaccinated children and their close contacts (vaccine-associated paralytic poliomyelitis or VAPP). OPV strains can circulate among susceptible individuals for long time in areas with absence of wild poliovirus transmission and suboptimal coverage with routine immunization resulting in low population immunity. Prolonged person-to-person transmission can result in genetic changes and the emergence of circulating vaccine-derived polioviruses (cVDPV) with neurovirulence and transmissibility characteristics of WPV. Type 2 poliovirus was responsible for about 40% of annual VAPP cases reported, and 85% paralytic cases caused by cVDPVs during 2000-2015. Based on SAGE recommendation this led to removal of type 2 by switching from tOPV to bOPV in primary immunization and introduction of "at least one dose of IPV in routine immunization" in most of the countries of the world.

Rationale for the study and expected outcomes and benefits for the GPEI

Several recent studies have demonstrated that, although a single dose would result in seroconversion to type 2 for a limited number of infants (32% to 80% depending on the age of administration and study), a high proportion (>90%) of those infants who are seronegative, may actually "primed" by that single dose. Although it is not clear whether priming may protect directly against paralysis if a type 2 cVDPV 2 outbreak emerges, primed children should develop protective antibody levels quickly following a new OPV or IPV dose provided as a response to the outbreak.

Studies assessing long-term immunity to IPV or OPV were conducted in individuals receiving three or more doses of poliovirus vaccines who could have been exposed to circulating wild or vaccine poliovirus. It is unknown whether the proportion of children who were seropositive or primed following a single dose of IPV will stay positive or primed, and for how long this immune response will persist. Additionally IPV delivered in clinics and outreach sites in low-resource countries may not produce the same response to those observed in clinical trials due to programmatic issues.

Furthermore, global shortage of IPV resulting in IPV stock out in many countries including Nepal led many children to miss out their IPV dose in routine immunization. Reliable estimates of population immunity in a country or region based upon coverage and estimated immunogenicity of the type of vaccine and vaccination schedules received, are crucial to guide programmatic decisions and manage vaccine supply for outbreak responses to type 2 poliovirus.

Therefore, a cross-sectional study is being conducted to determine whether the immune response provided by a single dose of IPV persists for more than a year, by assessing the proportion of children born after the tOPV-bOPV switch and vaccinated with a single dose of IPV at about 14 weeks in routine immunization who are still seropositive or primed at around two years of age. These new estimates will inform the GPEI on vaccine choices for responding to type 2 VDPV outbreaks and guide decisions on polio immunization schedules after cessation of all OPV types.

Objectives

The study primarily will compare the proportion of infants vaccinated with one dose of IPV after 14 weeks of age who are seropositive or primed against type 2 poliovirus, either > 21 months after vaccination (study group), or one month after vaccination (control group). Also we would determine the proportion of children seropositive to types 1 and 3 following a sequential bOPV-IPV or bOPV alone schedule, delivered through routine immunization services in a low resource country.

Study Design/ Procedures

This is an open-label phase IV clinical trial assessing immunogenicity to IPV. Study participants will be identified through screening of children who attend outpatient clinics at the study sites for well-child visits, immunization or minor illness. After screening, confirmation of eligibility and obtaining consent, children will be allocated to one of the two study arms, and given a dose of IPV after collecting clinical information and obtaining a blood sample. Children will be followed up according to the schedule for study arms to assess study objectives.

Blood sample will be centrifuged within 24 hours of collection, serum aliquoted into two cryovials and stored at Institute of Medicine (IOM) laboratory at -20*C until final shipment to Centers for Disease Control and Prevention(CDC), Atlanta. Determination of poliovirus antibodies will be conducted using a microneutralization testing. Titers below 1:8 will be considered negative and the highest detectable titer will be 1:1448.

Sample size and analytic plan:

The sample size will be powered to address the primary objective based on previous trials that have shown 90 - 100% of children to develop detectable immunity to type 2 poliovirus after IPV dose. Using a one-sided test for differences between proportions with a continuity correction Z-test using pooled variance (PASS v14), 237 children will be required in each group to detect a one-sided difference of ≥10% with 90% power and 0.05 alpha. To account for potential 5% drop-outs, the sample will be rounded up to 250 per group or 500 children total.

ELIGIBILITY:
Inclusion Criteria:

We will be including Nepali infants who fulfil the following criteria:

* Born after 30 April 2016
* Healthy infant or mild illness
* Age groups within one of the following age groups: 7-12 months or >24 months.
* Receipt of one dose of IPV at 3- 6 months of age (if age >24months) or zero doses (if age within 7-12 months). IPV receipt must be validated through immunization card or registry book.
* Parents that consent for participation in the full length of the study.
* Parents those are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute infection or illness at the time of enrollment that would require infant's admission to a hospital.
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Known allergy/sensitivity or reaction to polio vaccines.

Discontinuation Criteria

* Withdrawal of consent for participation for any reason.
* Request by parents of participant to terminate all study procedures.
* Identification of immunodeficiency disorder, bleeding disorder or another medical condition for which continued participation, in the opinion of the principal investigator, would pose a risk to the participant to continue in the study.
* Receipt of immunosuppressive medications.
* Receipt of any polio (OPV or IPV) vaccine outside of study after enrollment (as per parent's report).
* Allergic reaction to a dose of polio vaccine.
* Unable to collect or obtain blood at enrollment.
* Premature termination of the study.
* Temporary discontinuation of study activities may occur if there is a mOPV2 campaign.

Ages: 7 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of children with detectable immunity against type 2 poliovirus | 5 weeks
  To compare the proportion of infants vaccinated with one dose of IPV after 14 weeks of age who are seropositive or primed against type 2 poliovirus, either > 21 months after vaccination (study group), or one month after vaccination (control group)

SECONDARY OUTCOMES:
Proportion of children who seroconvert or boost antibody titers to type 2 poliovirus | 5 weeks
  To assess the proportion of children who seroconvert or boost antibody titers to type 2 poliovirus 30 days after a second dose of IPV, administered > 1 year after the first dose.

CONTACTS AND LOCATIONS:
Overall Officials: Laxman P Shrestha, MD, Principal Investigator — Tribhuvan University Teaching Hospital, Institute Of Medicine.; Concepcion Estivariz, MD, Principal Investigator — Centers for Disease Control and Prevention; Harish Verma, DCH, Principal Investigator — World Health Organization
Locations (3):
- Nepal (3):
  - Kanti Children's Hospital, Kathmandu
  - Patan Hospital, Kathmandu
  - Tribhuvan University Teaching Hospital, Kathmandu

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) sharing plan is undecided till now because the laboratory analysis is pending at CDC. IPD sharing plan will be revised after all results become available after agreement with collaborators in accordance to WHO and CDC guidelines

REFERENCES:
- [Background] Nathanson N, Kew OM. From emergence to eradication: the epidemiology of poliomyelitis deconstructed. Am J Epidemiol. 2010 Dec 1;172(11):1213-29. doi: 10.1093/aje/kwq320. Epub 2010 Oct 26. PMID 20978089
- [Background] Sutter RW, Kew OM, Cochi SL and Aylward RB. Poliovirus vaccine - live. In: Plotkin SA, Orenstein WA and Offit PA, eds. Vaccines. 6th ed: Elsevier, 2013:598-645
- [Background] Sutter RW, Patriarca PA. Inactivated and live, attenuated poliovirus vaccines: mucosal immunity. In: Kurstak E, ed. Measles and poliomyelitis. Austria: Springer-Verlag, 1993:279-293
- [Background] Vidor E, Plotkin SA. Poliovirus vaccine - Inactivated. In: Plotkin SA, Orenstein WA and Offit PA, eds. Vaccine. 6th ed. Philadelphia: Elsevier, 2013:573-597
- [Background] Roivainen M, Thoden CJ, Stenvik M, Poyry T, Hovi T. Virus excretion and strain specific antibody responses after oral poliovaccine in previously immunised children. J Med Virol. 1987 Nov;23(3):249-56. doi: 10.1002/jmv.1890230307. PMID 2828521
- [Background] Dowdle WR, Cochi SL. Global eradication of poliovirus: History and rationale. In: Semler BL, Wimmer E, eds. Molecular Biology of Picornaviruses. Washington: ASM Press, 2002:473-480
- [Background] Patriarca PA, Linkins RW and Sutter RW. Poliovirus vaccine formulations. In: Kurstak E, ed. Measles and Poliomyelitis. Wiena: Springer-Verlag, 1993:267-277
- [Background] Patriarca PA, Wright PF, John TJ. Factors affecting the immunogenicity of oral poliovirus vaccine in developing countries: review. Rev Infect Dis. 1991 Sep-Oct;13(5):926-39. doi: 10.1093/clinids/13.5.926. PMID 1660184
- [Background] Sutter RW, John TJ, Jain H, Agarkhedkar S, Ramanan PV, Verma H, Deshpande J, Singh AP, Sreevatsava M, Malankar P, Burton A, Chatterjee A, Jafari H, Aylward RB. Immunogenicity of bivalent types 1 and 3 oral poliovirus vaccine: a randomised, double-blind, controlled trial. Lancet. 2010 Nov 13;376(9753):1682-8. doi: 10.1016/S0140-6736(10)61230-5. Epub 2010 Oct 25. PMID 20980048
- [Background] Estivariz CF, Anand A, Gary HE Jr, Rahman M, Islam J, Bari TI, Wassilak SG, Chu SY, Weldon WC, Pallansch MA, Heffelfinger JD, Luby SP, Zaman K. Immunogenicity of three doses of bivalent, trivalent, or type 1 monovalent oral poliovirus vaccines with a 2 week interval between doses in Bangladesh: an open-label, non-inferiority, randomised, controlled trial. Lancet Infect Dis. 2015 Aug;15(8):898-904. doi: 10.1016/S1473-3099(15)00094-8. Epub 2015 Jun 17. PMID 26093980
- [Background] Estivariz CF, Pallansch MA, Anand A, Wassilak SG, Sutter RW, Wenger JD, Orenstein WA. Poliovirus vaccination options for achieving eradication and securing the endgame. Curr Opin Virol. 2013 Jun;3(3):309-15. doi: 10.1016/j.coviro.2013.05.007. Epub 2013 Jun 10. PMID 23759252
- [Background] Dayan GH, Thorley M, Yamamura Y, Rodriguez N, McLaughlin S, Torres LM, Seda A, Carbia M, Alexander LN, Caceres V, Pallansch MA. Serologic response to inactivated poliovirus vaccine: a randomized clinical trial comparing 2 vaccination schedules in Puerto Rico. J Infect Dis. 2007 Jan 1;195(1):12-20. doi: 10.1086/508427. Epub 2006 Nov 28. PMID 17152004
- [Background] Resik S, Tejeda A, Lago PM, Diaz M, Carmenates A, Sarmiento L, Alemani N, Galindo B, Burton A, Friede M, Landaverde M, Sutter RW. Randomized controlled clinical trial of fractional doses of inactivated poliovirus vaccine administered intradermally by needle-free device in Cuba. J Infect Dis. 2010 May 1;201(9):1344-52. doi: 10.1086/651611. PMID 20350164
- [Background] Mohammed AJ, AlAwaidy S, Bawikar S, Kurup PJ, Elamir E, Shaban MM, Sharif SM, van der Avoort HG, Pallansch MA, Malankar P, Burton A, Sreevatsava M, Sutter RW. Fractional doses of inactivated poliovirus vaccine in Oman. N Engl J Med. 2010 Jun 24;362(25):2351-9. doi: 10.1056/NEJMoa0909383. PMID 20573923
- [Background] Anand A, Zaman K, Estivariz CF, Yunus M, Gary HE, Weldon WC, Bari TI, Steven Oberste M, Wassilak SG, Luby SP, Heffelfinger JD, Pallansch MA. Early priming with inactivated poliovirus vaccine (IPV) and intradermal fractional dose IPV administered by a microneedle device: A randomized controlled trial. Vaccine. 2015 Nov 27;33(48):6816-22. doi: 10.1016/j.vaccine.2015.09.039. Epub 2015 Oct 23. PMID 26476367
- [Background] Ghendon Y, Robertson SE. Interrupting the transmission of wild polioviruses with vaccines: immunological considerations. Bull World Health Organ. 1994;72(6):973-83. PMID 7867144
- [Background] Sutter RW, Cochi SL and Melnick J. Poliovirus vaccine - live. 2002
- [Background] Ogra PL, Fishaut M, Gallagher MR. Viral vaccination via the mucosal routes. Rev Infect Dis. 1980 May-Jun;2(3):352-69. doi: 10.1093/clinids/2.3.352. PMID 6997965
- [Background] Ogra PL, Okayasu H, Czerkinsky C, Sutter RW. Mucosal immunity to poliovirus. Expert Rev Vaccines. 2011 Oct;10(10):1389-92. doi: 10.1586/erv.11.106. PMID 21988303
- [Background] Swartz TA, Handsher R, Stoeckel P, Drucker J, Caudrelier P, Van Wezel AL, Cohen H, Salk D, Salk J. Immunologic memory induced at birth by immunization with inactivated polio vaccine in a reduced schedule. Eur J Epidemiol. 1989 Jun;5(2):143-5. doi: 10.1007/BF00156819. PMID 2767220
- [Background] Resik S, Tejeda A, Sutter RW, Diaz M, Sarmiento L, Alemani N, Garcia G, Fonseca M, Hung LH, Kahn AL, Burton A, Landaverde JM, Aylward RB. Priming after a fractional dose of inactivated poliovirus vaccine. N Engl J Med. 2013 Jan 31;368(5):416-24. doi: 10.1056/NEJMoa1202541. PMID 23363495
- [Background] Asturias EJ, Bandyopadhyay AS, Self S, Rivera L, Saez-Llorens X, Lopez E, Melgar M, Gaensbauer JT, Weldon WC, Oberste MS, Borate BR, Gast C, Clemens R, Orenstein W, O'Ryan G M, Jimeno J, Clemens SA, Ward J, Ruttimann R; Latin American IPV001BMG Study Group. Humoral and intestinal immunity induced by new schedules of bivalent oral poliovirus vaccine and one or two doses of inactivated poliovirus vaccine in Latin American infants: an open-label randomised controlled trial. Lancet. 2016 Jul 9;388(10040):158-69. doi: 10.1016/S0140-6736(16)00703-0. Epub 2016 May 19. PMID 27212429
- [Background] Sutter RW, Bahl S, Deshpande JM, Verma H, Ahmad M, Venugopal P, Rao JV, Agarkhedkar S, Lalwani SK, Kunwar A, Sethi R, Takane M, Mohanty L, Chatterjee A, John TJ, Jafari H, Aylward RB. Immunogenicity of a new routine vaccination schedule for global poliomyelitis prevention: an open-label, randomised controlled trial. Lancet. 2015 Dec 12;386(10011):2413-21. doi: 10.1016/S0140-6736(15)00237-8. Epub 2015 Sep 18. PMID 26388534
- [Background] Carlsson RM, Claesson BA, Fagerlund E, Knutsson N, Lundin C. Antibody persistence in five-year-old children who received a pentavalent combination vaccine in infancy. Pediatr Infect Dis J. 2002 Jun;21(6):535-41. doi: 10.1097/00006454-200206000-00011. PMID 12182378
- [Background] McBean AM, Thoms ML, Albrecht P, Cuthie JC, Bernier R. Serologic response to oral polio vaccine and enhanced-potency inactivated polio vaccines. Am J Epidemiol. 1988 Sep;128(3):615-28. doi: 10.1093/oxfordjournals.aje.a115009. PMID 2843039
- [Background] Halperin SA, Smith B, Russell M, Scheifele D, Mills E, Hasselback P, Pim C, Meekison W, Parker R, Lavigne P, Barreto L. Adult formulation of a five component acellular pertussis vaccine combined with diphtheria and tetanus toxoids and inactivated poliovirus vaccine is safe and immunogenic in adolescents and adults. Pediatr Infect Dis J. 2000 Apr;19(4):276-83. doi: 10.1097/00006454-200004000-00003. PMID 10783014
- [Background] Zimmermann U, Gavazzi G, Richard P, Eymin C, Soubeyrand B, Baudin M. Immunogenicity and safety of a booster dose of diphtheria, tetanus, acellular pertussis and inactivated poliomyelitis vaccine (Tdap-IPV; Repevax) administered concomitantly versus non-concomitantly with an influenza vaccine (Vaxigrip) to adults aged >/=60 years: an open-label, randomised trial. Vaccine. 2013 Mar 1;31(11):1496-502. doi: 10.1016/j.vaccine.2012.12.081. Epub 2013 Jan 10. PMID 23313654
- [Background] Abbink F, Buisman AM, Doornbos G, Woldman J, Kimman TG, Conyn-van Spaendonck MA. Poliovirus-specific memory immunity in seronegative elderly people does not protect against virus excretion. J Infect Dis. 2005 Mar 15;191(6):990-9. doi: 10.1086/427810. Epub 2005 Feb 10. PMID 15717277
- [Background] Rumke HC, Oostvogel PM, Van Steenis G, Van Loon AM. Poliomyelitis in The Netherlands: a review of population immunity and exposure between the epidemics in 1978 and 1992. Epidemiol Infect. 1995 Oct;115(2):289-98. doi: 10.1017/s0950268800058416. PMID 7589268
- [Background] Kaml M, Weiskirchner I, Keller M, Luft T, Hoster E, Hasford J, Young L, Bartlett B, Neuner C, Fischer KH, Neuman B, Wurzner R, Grubeck-Loebenstein B. Booster vaccination in the elderly: their success depends on the vaccine type applied earlier in life as well as on pre-vaccination antibody titers. Vaccine. 2006 Nov 17;24(47-48):6808-11. doi: 10.1016/j.vaccine.2006.06.037. Epub 2006 Jul 10. PMID 16872725
- [Background] Estivariz CF, Jafari H, Sutter RW, John TJ, Jain V, Agarwal A, Verma H, Pallansch MA, Singh AP, Guirguis S, Awale J, Burton A, Bahl S, Chatterjee A, Aylward RB. Immunogenicity of supplemental doses of poliovirus vaccine for children aged 6-9 months in Moradabad, India: a community-based, randomised controlled trial. Lancet Infect Dis. 2012 Feb;12(2):128-35. doi: 10.1016/S1473-3099(11)70190-6. Epub 2011 Nov 7. PMID 22071249
- [Background] Moriniere BJ, van Loon FP, Rhodes PH, Klein-Zabban ML, Frank-Senat B, Herrington JE, Pallansch MA, Patriarca PA. Immunogenicity of a supplemental dose of oral versus inactivated poliovirus vaccine. Lancet. 1993 Jun 19;341(8860):1545-50. doi: 10.1016/0140-6736(93)90693-b. PMID 8099637
- [Background] Platt LR, Estivariz CF, Sutter RW. Vaccine-associated paralytic poliomyelitis: a review of the epidemiology and estimation of the global burden. J Infect Dis. 2014 Nov 1;210 Suppl 1(Suppl 1):S380-9. doi: 10.1093/infdis/jiu184. PMID 25316859
- [Background] Burns CC, Diop OM, Sutter RW, Kew OM. Vaccine-derived polioviruses. J Infect Dis. 2014 Nov 1;210 Suppl 1:S283-93. doi: 10.1093/infdis/jiu295. PMID 25316847
- [Background] Kew OM, Sutter RW, de Gourville EM, Dowdle WR, Pallansch MA. Vaccine-derived polioviruses and the endgame strategy for global polio eradication. Annu Rev Microbiol. 2005;59:587-635. doi: 10.1146/annurev.micro.58.030603.123625. PMID 16153180
- [Background] Meeting of the Strategic Advisory Group of Experts on Immunization, November 2012 - conclusions and recommendations. Wkly Epidemiol Rec. 2013 Jan 4;88(1):1-16. No abstract available. English, French. PMID 23311010
- [Background] Tebbens RJ, Pallansch MA, Kew OM, Caceres VM, Jafari H, Cochi SL, Sutter RW, Aylward RB, Thompson KM. Risks of paralytic disease due to wild or vaccine-derived poliovirus after eradication. Risk Anal. 2006 Dec;26(6):1471-505. doi: 10.1111/j.1539-6924.2006.00827.x. PMID 17184393
- [Background] Thompson KM, Duintjer Tebbens RJ. National choices related to inactivated poliovirus vaccine, innovation and the endgame of global polio eradication. Expert Rev Vaccines. 2014 Feb;13(2):221-34. doi: 10.1586/14760584.2014.864563. Epub 2013 Dec 4. PMID 24308581
- [Background] O'Ryan M, Bandyopadhyay AS, Villena R, Espinoza M, Novoa J, Weldon WC, Oberste MS, Self S, Borate BR, Asturias EJ, Clemens R, Orenstein W, Jimeno J, Ruttimann R, Costa Clemens SA; Chilean IPV/bOPV study group. Inactivated poliovirus vaccine given alone or in a sequential schedule with bivalent oral poliovirus vaccine in Chilean infants: a randomised, controlled, open-label, phase 4, non-inferiority study. Lancet Infect Dis. 2015 Nov;15(11):1273-82. doi: 10.1016/S1473-3099(15)00219-4. Epub 2015 Aug 26. PMID 26318714
- [Derived] Sharma AK, Verma H, Estivariz CF, Bajracharaya L, Rai G, Shah G, Sherchand J, Jones KAV, Mainou BA, Chavan S, Jeyaseelan V, Sutter RW, Shrestha LP. Persistence of immunity following a single dose of inactivated poliovirus vaccine: a phase 4, open label, non-randomised clinical trial. Lancet Microbe. 2023 Nov;4(11):e923-e930. doi: 10.1016/S2666-5247(23)00215-X. Epub 2023 Sep 26. PMID 37774729
- See also: Global Polio Eradication Initiative. List of wild poliovirus by country and year. — http://polioeradication.org/polio-today/polio-now/wild-poliovirus-list
- See also: The Global Polio Eradication Initiative. Data and monitoring — http://www.polioeradication.org
- See also: Hickling J, Jones R and Nundy N. Improving the affordability of intactivated poliovirus vaccine (IPV) for use in low-and middle-income countries — http://www.path.org
- See also: Global Polio Eradication Initiative. Standard Operating Procedures: responding to a poliovirus event and outbreak, part 2: protocol for poliovirus type 2, 15 August 2016 (Original publication 20 april 2016) — http://polioeradication.org/tools-and-library/resources-for-polio-eradicators/gpei-tools-protocols-and-guidelines/
- See also: Department of Immunization Vaccines and Biologicals. WHO multi-dose vial policy (MDVP), Revision 2014. WHO/IVB/14.07 — http://apps.who.int/iris/bitstream/10665/135972/1/WHO_IVB_14.07_eng.pdf